CLINICAL TRIAL: NCT00964990
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-42160443 in Subjects With Postherpetic Neuralgia and Post-traumatic Neuralgia, Followed by a Double Blind Safety Extension and an Open-label Safety Extension
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-42160443 in Patients With Neuropathic Pain (Postherpetic Neuralgia and Post-traumatic Neuralgia)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistic reasons associated with the FDA-imposed clinical hold.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR016474; 42160443NPP2001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); 2008-007478-39 (EudraCT Number)
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Pain; Neuralgia, Postherpetic; Neuralgia; Mononeuropathies
Keywords: Moderate to severe chronic peripheral neuropathic pain; Postherpetic neuralgia; Post-traumatic neuralgia; Moderate to severe chronic pain; JNJ-42160443
MeSH Terms: conditions — Pain; Neuralgia, Postherpetic; Neuralgia; Mononeuropathies | interventions — fulranumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 001 (Experimental): JNJ-42160443 SC injection (1 3 or 10 milligrams) once every 28 days
  Interventions: Drug: JNJ-42160443
- 002 (Placebo Comparator): Placebo SC injection once every 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42160443 — Type=exact number, unit=mg, number= 1, 3, or 10, form=solution for injection, route=Subcutaneous use. One injection of 1, 3, or 10 mg of JNJ-42160443 every 28 days for up to 52 wks and then every 4, 8, or 12 weeks for up to an additional 52 weeks
  Arms: 001
Drug: Placebo — Form=solution for injection, route=Subcutaneous injection. One injection of matching placebo every 28 days for up to 52 wks
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of JNJ-42160443 in the treatment of moderate to severe neuropathic pain in patients with a diagnosis of postherpetic neuralgia and post-traumatic neuralgia.

DETAILED DESCRIPTION:
The current study is a randomized (study drug assigned by chance), double-blind (neither the study doctor nor the patient knows the name of the assigned drug), placebo-controlled, dose-ranging study to evaluate the efficacy, safety, and tolerability of JNJ-42160443 in patients with postherpetic neuralgia and post-traumatic neuralgia, followed by a double blind extension and an open-label (study doctor and patient knows the name of the study drug) extension. This study will evaluate the safety and effectiveness of JNJ-42160443 in the treatment of patients with moderate to severe, chronic, neuropathic pain that is not controlled with or without standard pain therapy and who have a diagnosis of postherpetic neuralgia (PHN) or post-traumatic neuralgia. The total duration of the study will be approximately 130 weeks (i.e., includes screening phase, 12-week double-blind efficacy phase, double-blind safety extension phase, and the open-label safety extension phase). During the 12 week treatment and 40 week double-blind extension phases, PHN patients will receive Placebo, JNJ 42160443 1, 3, or 10 mg and post-traumatic neuralgia patients will receive placebo or JNJ-42160443 10 mg; all doses will be given as a single, subcutaneous (under the skin) (SC) injection every 28 days. During the 52-week open-label extension phase, all patients will receive a single SC injection of JNJ-42160443 up to 10 mg every 4, 8, or 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with postherpetic neuralgia or post-traumatic neuralgia and who have chronic neuropathic pain (pain persistent for > 6 months) that is moderate to severe; Currently taking pain medication but are not adequately controlled by standard of care or are not currently taking pain medications because intolerable to, or not willing to use, standard of care. Exclusion Criteria: History of a separate pain condition (e.g., joint osteoarthritis) that is more severe than pain due to diagnosis of PHN or post-traumatic neuralgia

* Patients with post-traumatic neuralgia that are characteristic of complex regional pain syndrome Type I
* Patients with lumbar-sacral radiculopathy, failed low-back surgery, or spinal cord injury
* Patient whose nerve injury or pain is expected to recover in the next 4 months
* Patients with evidence of another neuropathic pain not under study, such as pain resulting from diabetic painful neuropathy, sensory neuropathies or pain caused by radiation, chemotherapy, alcohol, HIV infection
* Other peripheral neuropathy, paresthesia, or dysesthesia, or any other previously diagnosed neurologic condition causing the above noted symptoms that is not related with the PHN or post-traumatic neuralgia under the study
* Women who are pregnantHistory of a separate pain condition (e.g., joint osteoarthritis) that is more severe than pain due to diagnosis of PHN or post-traumatic neuralgia; Patients with post-traumatic neuralgia that are characteristic of complex regional pain syndrome Type I; Patients with lumbar-sacral radiculopathy, failed low-back surgery, or spinal cord injury; Patient whose nerve injury or pain is expected to recover in the next 4 months; Patients with evidence of another neuropathic pain not under study, such as pain resulting from diabetic painful neuropathy, sensory neuropathies or pain caused by radiation, chemotherapy, alcohol, HIV infection; Other peripheral neuropathy, paresthesia, or dysesthesia, or any other previously diagnosed neurologic condition causing the above noted symptoms that is not related with the PHN or post-traumatic neuralgia under the study; Women who are pregnant or breast-feeding; Type I or Type II diabetes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The daily evening assessment of average pain intensity | Baseline (7 days before randomization) and last 7 days of the 12-week treatment phase

SECONDARY OUTCOMES:
Pain at its worst | Daily for 12 weeks
Brief Pain Inventory | Up to Week 13 (ie, at Visits 1, 3, 7, 8, 9)
Neuropathic pain symptom inventory | Up to Week 13 (ie, at Visits 1, 3, 7, 8, 9)
Patient Global Impression of Change | Up to Week 13 (ie, at Visits 1, 3, 7, 8, 9)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (48):
- United States (40):
  - Tucson, Arizona
  - Fresno, California
  - Redondo Beach, California
  - Roseville, California
  - Hollywood, Florida
  - Oldsmar, Florida
  - Palm Beach Gardens, Florida
  - Port Orange, Florida
  - St. Petersburg, Florida
  - Sunrise, Florida
  - Tamarac, Florida
  - Decatur, Georgia
  - Boise, Idaho
  - Lewiston, Idaho
  - Evansville, Indiana
  - Franklin, Indiana
  - Lexington, Kentucky
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Brockton, Massachusetts
  - Hyannis, Massachusetts
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Meridian, New Jersey
  - Albany, New York
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Allentown, Pennsylvania
  - Altoona, Pennsylvania
  - Pennsburg, Pennsylvania
  - Philadelphia, Pennsylvania
  - Greer, South Carolina
  - Nashville, Tennessee
  - Smyrna, Tennessee
  - Dallas, Texas
  - Plano, Texas
  - San Antonio, Texas
- Belgium (3):
  - Edegem
  - Leuven
  - Waterschei-Zwartberg
- Netherlands (2):
  - Alkmaar
  - Maastricht
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia

REFERENCES:
- [Derived] Wang H, Romano G, Fedgchin M, Russell L, Sanga P, Kelly KM, Frustaci ME, Thipphawong J. Fulranumab in Patients With Pain Associated With Postherpetic Neuralgia and Postraumatic Neuropathy: Efficacy, Safety, and Tolerability Results From a Randomized, Double-blind, Placebo-controlled, Phase-2 Study. Clin J Pain. 2017 Feb;33(2):99-108. doi: 10.1097/AJP.0000000000000388. PMID 27153360